CLINICAL TRIAL: NCT06185595
Title: Effect of Glycerol-Electrolyte Beverages on Fluid Balance in Healthy Euhydrated Men and Women at Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2311
Record Dates: First submitted 2023-12-08; First posted 2023-12-29 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Hydration
Keywords: hydration; euhydration; fluid balance; fluid retention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (Placebo Comparator): No sodium, No glycerol
  Interventions: Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order.
- Sodium only group 1 (Experimental): 55 mmol/L sodium
  Interventions: Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order.
- Glycerol only (Experimental): 4.6% glycerol
  Interventions: Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order.
- Sodium and Glycerol group 1 (Experimental): 55 mmol/L sodium and 4.6% glycerol
  Interventions: Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order.
- Sodium only group 2 (Experimental): 27.5 mmol/L sodium
  Interventions: Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order.
- Sodium and Glycerol group 2 (Experimental): 27.5 mmol/L sodium and 2.3% glycerol
  Interventions: Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order.

INTERVENTIONS:
Other: Beverage. Incomplete block where each participant will complete 3 of the 6 possible glycerol-sodium blends in random order. — 9.3 oz (273 ml) aliquot of one of the study beverages every 15 min for a total of 28 oz (828 ml) over a 45-min period, followed by 15 min of rest. Flavored water matched for sweetness, color. flavor, but cannot be matched for saltiness. All sodium-containing drinks will include a base blend of other electrolytes (potassium 15 mmol/L, magnesium 8 mmol/L, and calcium 5 mmol/L).

SUMMARY:
The objective of this study is to determine the effect of consumption of drinks with varying amounts of glycerol and electrolytes on fluid balance at rest.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* If female, subject is not pregnant
* Subject is 18-50 years of age, inclusive
* You are at least recreationally active (engaged in light to moderate-intensity, intermittent, or steady-state exercise at least 3 days per week for at least 30 min at a time)
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study (e.g., diuretics)
* Subject has no health conditions that would interfere with the study as indicated on the general health questionnaire (GHQ), e.g. cardiovascular, renal, or metabolic diseases
* Subject is willing to avoid alcohol consumption 24 hours prior to visit(s)
* Subject is willing to fast overnight (~8-12 hours)
* Subject is willing to refrain from vigorous exercise for 24 hours
* Subject is willing to eat the exact same food the day prior to each visit to the laboratory
* Able to speak, write, and read English
* Provision of written consent to participate

Exclusion Criteria:

* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Fluid balance | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90,120 and 180 minutes
  Change in body mass to the nearest 0.005 kilogram (kg) using a platform scale

SECONDARY OUTCOMES:
Fluid retention | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90,120 and 180 minutes
  As a percent (%)
Urine mass | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90, 120 and 180 minutes
  By urine mass scale in grams (g)
Urine specific gravity | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90,120 and 180 minutes
  By USG digital pen refractometer
Blood sodium | Change from baseline (pre-beverage) to post-beverage Time 0, 60 min, 120 min and 180 minutes
  By iSTAT Blood Electrolyte and Chemistry Analyzer (CG8+ cartridge) in mmol/L
Blood glucose | Screening visit only
  Glucometer for point of care test in mg/dL
Blood glucose | Change from baseline (pre-beverage) to post-beverage Time 0, 60 min, 120 min and 180 minutes
  By iSTAT Blood Electrolyte and Chemistry Analyzer (CG8+ cartridge) in mg/dL
Percent change in plasma volume | Change from baseline (pre-beverage) to post-beverage Time 0, 60 min, 120 min and 180 minutes
  Calculated from hematocrit and hemoglobin concentration
Serum glycerol concentration | Change from baseline (pre-beverage) to post-beverage Time 0, 60 min, 120 min and 180 minutes
  By Sigma Aldrich glycerol assay kit in mmol/L
Blood pressure | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90, 120 and 180 minutes
  mmHg by automatic sphygmomanometer
Heart rate | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90, 120 and 180 minutes
  Beats per minute (bpm) by heart rate monitor
Subjective measures of gastrointestinal discomfort and headache | Change from baseline (pre-beverage) to post-beverage Time 0, 30, 60, 90, 120 and 180 minutes
  Visual Analog Scale (VAS) symptom rating of how you feel right now by placing a slash along a 100 millimeter (mm) vertical line anchored from 0 mm (None) to 100 mm (Severe). Fewer symptoms and lower numbers are better.
Menstrual cycle phase | Female participants log menstrual flow throughout study participation. The three study sessions (2-45 days apart) are scheduled to avoid menses and can be completed in the same menstrual cycle, or in 3 different cycles (3 different months) if needed.
  Date of last menstrual period by self-report of female participant

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Principal Investigator — PepsiCo, Inc. Sports Science
Locations (1):
- PepsiCo R&D, Gatorade Sports Science Institute, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker LB, Hinkley JM, Ozga M, Alfred SL, Merritt JR, De Chavez PJD. A randomized trial modeling the effects of solutions with low to moderate glycerol and sodium concentrations on fluid balance in healthy, active adults. Am J Clin Nutr. 2026 Jan;123(1):101094. doi: 10.1016/j.ajcnut.2025.10.011. Epub 2025 Oct 23. PMID 41138915